CLINICAL TRIAL: NCT03693547
Title: Open, Multicenter, Monotherapy, Phase II Clinical Study of Utidelone Injection in Patients With Advanced Non-small Cell Lung Cancer After Failure or Intolerability to Second-line Standard Treatment
Brief Title: Clinical Study of Utidelone Injection in Patients With Advanced Non-small Cell Lung Cancer（NSCLC）
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Chengdu Biostar Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG01-1801
Record Dates: First submitted 2018-09-29; First posted 2018-10-03 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- utidelone (Experimental): Utidelone Injection: 30 mg/m2/day, IV on day 1-day 5 of each 21 day cycle, administered to enrolled patients with advanced NSCLC
  Interventions: Drug: utidelone injection

INTERVENTIONS:
Drug: utidelone injection — utidelone monotherapy in patients with advanced NSCLC by utidelone
  Other Names: UTD1 injection

SUMMARY:
To assess the effectiveness and safety of utidelone injection in patients with advanced or metastatic NSCLC as a phase II trial

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung cancer
2. NSCLC patients who are not suitable for surgery or radical radiotherapy or chemotherapy, or who have failed to or are intolerable for standard treatment in local advanced or metastatic NSCLC;
3. NSCLC patients failed or intolerable to previous standard second-line treatment (including platinum chemotherapy or targeted therapy);
4. Patients who did not receive chemotherapy, radiotherapy, surgical therapy, molecularly targeted drug therapy, or immunotherapy 4 weeks prior to enrollment;
5. Age 18 -70 years old, ECOG performance status of 0-1; Life expectancy of 3 months or more;
6. Patients must have measurable disease, defined as at least one target lesion that can be accurately measured by imaging techniques in at least one dimension as ≥20 mm with conventional computed tomography (CT), ≥10 mm with spiral CT scan (≥15mm for lymph node) within 3 weeks before enrolment;
7. Patients with no brain metastases or with brain metastases but are stable for more than 4 weeks after treatment;
8. Peripheral neuropathy (PN) <grade 2 on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 within 4 weeks before enrolment;
9. Patients must have normal haematology as defined below: HGB ≥9 g/L, absolute neutrophil count ≥1.5×109/L, platelets ≥80×109/L, bilirubin ≤1.5× the upper limit of normal (ULN) (patients with liver metastasis ≤3xULN), aspartate transaminase (AST)/ alanine transaminase (ALT) ≤2.5 ×ULN (patients with liver metastasis ≤5xULN), and creatinine clearance ≥45 mL/min;
10. Patients with no major organ dysfunctions and heart disease;
11. Patients who give written informed consent with good compliance.

Exclusion Criteria:

1. Patients who are pregnant or breast feeding;
2. Patients with active tuberculosis
3. Patients with high possibility of interstitial lung disease ;
4. Patients with comorbidities, such as carcinomatous meningitis, central nervous system (CNS) metastasis, other active malignancies requiring simultaneous treatment, but not including cervical cancer in situ or basal cell carcinoma of the skin, severe disorders of the heart, lung, liver, or kidneys, severe hypertension, uncontrolled diabetes, severe gastrointestinal ulceration, active infections in need of antibiotics, or with incontrollable psychiatric history;
5. patients with HIV, untreated active hepatitis；
6. Patients with poor compliance;
7. Patients not fitted for this study determined by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Tumor response to utidelone treatment | 6 months from first study treatment
  Reflected by percentage of tumor size reduction or regression, assessed by imaging techniques and expressed as Objective Response Rate (ORR）ORR is defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) according to RECIST. 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 1 year from first study treatment
  PFS is defined as the duration of time from first study treatment to disease progression or death from any cause as documented by the investigator
Overall survival (OS) | 2 year from enrolment
  OS is defined as the duration of time from first study treatment until death from any cause.
Incidence of treatment-emergent adverse events based the Common Terminology Criteria for Adverse Events (CTCAE) version 4·03 | 1 year from first study treatment
  Observe and record incidence of adverse events and severe adverse events associated with utidelone treatment, assessed by investigators according to CTCAE version 4·03

CONTACTS AND LOCATIONS:
Overall Officials: YUANKAI SHI, MD, PhD, Principal Investigator — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China
Locations (4):
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Shi Y, Chen G, Zhao Y, Zhao J, Lin L. Efficacy and safety of utidelone for the treatment of patients with locally advanced or metastatic non-small-cell lung cancer who have failed standard second-line treatment: A phase 2 clinical trial (BG01-1801). Cancer Pathog Ther. 2023 Oct 29;2(2):103-111. doi: 10.1016/j.cpt.2023.10.006. eCollection 2024 Apr. PMID 38601485